CLINICAL TRIAL: NCT01688947
Title: A Phase 2, Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group, Multicenter Study Evaluating the Analgesic Efficacy and Safety of V116517 in Subjects With Moderate to Severe Chronic Pain Due to Postherpetic Neuralgia (PHN)
Brief Title: Analgesic Efficacy and Safety of V116517 in Subjects With Moderate to Severe Chronic Pain Due to Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VND2002
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Postherpetic Neuralgia; Pain
Keywords: Pain; Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain | interventions — 4-(3-chloro-5-(1,2-dihydroxyethyl)-2-pyridyl)-N-(5-(trifluoromethyl)-2-pyridyl)-3,6-dihydro-2H-pyridine-1-carboxamide; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- V116517 - 50 mg (Experimental): V116517 50-mg tablets
  Interventions: Drug: V116517 50-mg tablets; Drug: Placebo
- V116517 - 30 mg (Experimental): V116517 30-mg tablets
  Interventions: Drug: V116517 30-mg tablets; Drug: Placebo
- Pregabalin (Active Comparator): Pregabalin capsules
  Interventions: Drug: Pregabalin capsules; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V116517 50-mg tablets — Taken orally twice daily
  Arms: V116517 - 50 mg
Drug: V116517 30-mg tablets — Taken orally twice daily
  Arms: V116517 - 30 mg
Drug: Pregabalin capsules — 1-2 capsules taken orally twice daily
  Arms: Pregabalin
Drug: Placebo — Tablets to match V116517 taken orally twice daily and/or placebo capsules to match pregabalin, 1-2 capsules taken orally twice daily

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of 2 dose levels of V116517 versus placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects with chronic pain due to PHN as their primary pain condition and some degree of pain every day from this condition.
2. Clinical diagnosis of PHN based on history of painful dermatomal blistering rash resolving in a few weeks followed by persistent pain in the same region of ≥ 3 months duration.

Key Exclusion Criteria:

1. Subjects with chronic pain conditions other than PHN as their predominant pain condition, including gout, pseudo gout, psoriatic arthritis, active Lyme disease, rheumatoid arthritis or any other inflammatory arthritis, fibromyalgia, neuropathic pain conditions, bursitis, or acute injury or signs of active infection in the target pain area.
2. Subjects who cannot or will not agree to stop all concomitant analgesic medications apart from specified protocol supplemental analgesic medications.
3. Subjects with a recent history of seizure within the past 5 years.
4. Subjects who use opioids more than 4 days per week.
5. Subjects with clinically unstable medical conditions, including cardiac disease (unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, or active myocardial ischemia); respiratory disease; biliary tract disease; hypothyroidism; adrenal cortical insufficiency; or any other medical condition that in the investigator's opinion is inadequately treated and precludes entry into the study.
6. Subjects with a history of suicide attempts, or subjects clinically judged by the principal investigator (PI) to be at serious risk of suicide.
7. PHN-pain-condition-specific exclusions:

   * Subjects who received pain-control interventions including neurolytic blocks or neurosurgical procedures to the affected nerve or spinal cord segment, spinal cord, stimulators, or neuraxial infusion pumps.
8. Active-comparator-related exclusions:

   * Subjects who are allergic to or cannot tolerate pregabalin or acetaminophen.

Other protocol specific inclusion/exclusion criteria may apply.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
"Pain on the average in the last 24 hours" score from the Modified Brief Pain Inventory - Short Form (mBPI-SF) | Week 4

SECONDARY OUTCOMES:
mBPI-SF severity of pain (parameters including average pain, worst pain, least pain, pain right now) and interference of pain (all parts of question 6) | Week 4
Neuropathic Pain Symptom Inventory (NPSI) | Week 4
Patient Global Impression of Change (PGIC) | Week 4
Supplemental Analgesic Medication Use | Over 4 weeks

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Investigational Site, Tucson, Arizona
  - Investigational Site, La Jolla, California
  - Investigational Site, North Hollywood, California
  - Investigational Site, Boca Raton, Florida
  - Investigational Site, Bradenton, Florida
  - Investigational Site, DeLand, Florida
  - Investigational Site, Fort Myers, Florida
  - Investigational Site, Lynn Haven, Florida
  - Investigational Site, North Miami, Florida
  - Investigational Site, Orlando, Florida
  - Investigational Site, Oviedo, Florida
  - Investigational Site, Palm Beach Gardens, Florida
  - Investigational Site, Sarasota, Florida
  - Investigational Site, St. Petersburg, Florida
  - Investigational Site, Sunrise, Florida
  - Investigational Site, Decatur, Georgia
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Prairie Village, Kansas
  - Investigational Site, New Bedford, Massachusetts
  - Investigational Site, Bay City, Michigan
  - Investigational Site, Bingham Farms, Michigan
  - Investigational Site, Pinconning, Michigan
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, Albuquerque, New Mexico
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Raleigh, North Carolina
  - Investigational Site, Austin, Texas
  - Investigational Site, Salt Lake City, Utah